CLINICAL TRIAL: NCT02537210
Title: Oral 5-aminosalicylic Acid Withdrawal in Long Standing Inactive Ulcerative Colitis: A Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Aminosalicylic Acid Withdrawal Study in Long Standing Inactive Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Queen Elizabeth Hospital, Hong Kong (Other); Alice Ho Miu Ling Nethersole Hospital (Other); Tseung Kwan O Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASA withdrawal study
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Colitis, Ulcerative; Aminosalicylic Acid
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesalazine (Active Comparator): mesalazine 2g od po for 12 months
  Interventions: Drug: Mesalazine
- Placebo oral capsule (Placebo Comparator): placebo 5 capsules od po for 12 months
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Mesalazine — Patients will be prescribed Asacol 2g daily for 12 months
  Other Names: Asacol
  Arms: Mesalazine
Drug: Placebo oral capsule — Patients will be prescribed placebo 5 capsules daily for 12 months
  Other Names: Placebo
  Arms: Placebo oral capsule

SUMMARY:
The purpose of this study is to determine whether aminosalicylic acid (ASA) can be safely withdrawn in patients with long-standing clinical inactive UC.

DETAILED DESCRIPTION:
This is a randomized, double-blind, controlled trial in which patients with long-standing clinically inactive UC receiving ASA for maintenance of remission will be randomized to either continue 5-ASA or to receive an equivalent placebo for 12 months. The primary endpoint is clinical relapse at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* have a confirmed diagnosis of UC according to established clinical, endoscopic and histologic criteria
* in long-standing clinical remission
* written informed consent

Exclusion Criteria:

* allergic to mesalazine
* prior bowel surgery except appendectomy
* hepatic or renal dysfunction
* malignant disease within 5 years
* pregnancy or breast feeding or women of child-bearing age without regular use of contraception
* on anti-tumor necrosis factor therapy
* terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
The differences of relapse rates between the two arms | 12 months
  Relapse rate of patient in both arms will be calculated

SECONDARY OUTCOMES:
Patients' drug compliance | 12 months
  Proportion of patients with good drug compliance, defined as more than 80% of drug taken will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Siew Ng, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No